CLINICAL TRIAL: NCT05139381
Title: Open Label, Observational Study for Children & Adolescent With Severe Asthma With an Eosinophilic Phenotype Treated With Mepolizumab
Brief Title: Study for Children & Adolescent With Severe Asthma With an Eosinophilic Phenotype Treated With Mepolizumab
Acronym: CASAM
Status: Active, not recruiting | Type: Observational
Sponsor: King's College Hospital NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 306475
Record Dates: First submitted 2021-11-17; First posted 2021-12-01 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Asthma in Children
MeSH Terms: interventions — mepolizumab

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Treated with Mepolizumab
  Interventions: Drug: Mepolizumab

INTERVENTIONS:
Drug: Mepolizumab — Treatment with Mepoluzimab

SUMMARY:
Open label, observational cohort study conducted to collect demographics, clinical characteristics and outcome observational data from children (6-17 years) with a clinical diagnosis of severe asthma in 2 countries (Spain and United Kingdom), in public institutions.

All eligible participants who have a physician decision to initiate mepolizumab treatment and are consented for the study will be observed.

Subjects must have received mepolizumab (Nucala) since authorisation by EMEA in September 2018 (in Spain since December 2019) as an add-on treatment for severe refractory eosinophilic asthma in paediatric patients aged six up to 17 years. The study will be implemented in 16 investigating sites (10 in Spain and 6 in UK). The assignment of a patient to a particular therapeutic strategy is not decided in advance by the study protocol, but is determined by the usual practice of medicine, and the decision to prescribe a particular drug is clearly dissociated from the decision to include the patient in the study.

Eligible participants will meet the local reimbursement criteria. The study will be managed by IQVIA. No patient-identifying information will be transferred to the sponsor nor the CRO.

No visits should be scheduled specifically for this observational study, data will be collected at usual asthma healthcare visits (routine or unscheduled, remote or face to face). If a participant is seen by their physician for monthly mepolizumab injections, data for healthcare utilization, asthma medications and any recent lung function assessment will be collected on a monthly basis. When the participant is seen less frequently by their physician (for example when mepolizumab injection is given at a different site or at home) this data will be collected at usual asthma healthcare visits, which are likely to occur less frequently.

The index date will be defined as the date of the first mepolizumab injection administration during the study (i.e. treatment initiation). To accommodate local healthcare practice, this will be according to local healthcare practice.

ELIGIBILITY:
Inclusion Criteria:

1. Patient who provides his/her written informed Consent to participate prior to commencing any study related activities.
2. Children & Adolescent aged 6-17 years at mepolizumab initiation
3. Patient with a current clinical diagnosis of severe asthma (as per GINA / ATS / ERS / BTS criteria) and eosinophilic phenotype (as per mepolizumab licence) at mepolizumab initiation
4. Patient currently under treatment or who initiates treatment with mepolizumab at the inclusion visit based on national asthma guidelines.
5. Patient with relevant paper or electronic-based medical records available for 12-months prior to enrolment date/ index date (date of first mepolizumab injection) for clinically significant asthma exacerbation.

Exclusion Criteria:

* A participant will not be eligible for inclusion in this study if any of the following criteria apply: 3. Patient who does not meet the inclusion criteria. 4. Patient who has participated in an asthma monoclonal antibodies drug interventional clinical trial in the previous 12-months to mepolizumab initiation.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: 100 paediatric patients (50 per country) using mepolizumab at severe asthma centres in the United Kingdom and Spain over 24-36 months.
Sampling Method: Probability Sample
Enrollment: 148 (Actual)
Dates: Start 2022-03-02 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03-12 (Estimated)

PRIMARY OUTCOMES:
To compare the rates of clinically significant asthma exacerbations in the pre-exposure and the 12-month post-exposure period with mepolizumab treatment. | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- King's College Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Gupta A, de Mir Messa I, Valverde-Molina J, Murray CS, Moral L, Torres Borrego J, Pike K, Diaz-Izquierdo A, Martinez-Canavate A, Nagakumar P, Cook J, Gupta L; CASAM Group. Protocol for an open labelled observational study in children & adolescents with severe asthma with an eosinophilic phenotype treated with mepolizumab (CASAM). PLoS One. 2025 Dec 19;20(12):e0335399. doi: 10.1371/journal.pone.0335399. eCollection 2025. PMID 41417800